CLINICAL TRIAL: NCT05365828
Title: Legacies and Futures: Gestational Parents' Experiences With Vulnerability and Resilience as it Influence Parent and Neonatal Health
Brief Title: Legacies and Futures: Measuring Roles of Resilience and Vulnerability in Pregnancy and Birth Outcomes
Status: Active, not recruiting | Type: Observational
Sponsor: University College, London (Other)
Collaborators: UCL, Bloomsbury and East London (UBEL) Doctoral Training Partnership (Unknown); Economic and Social Research Council, United Kingdom (Other); University College London Hospitals (Other); King's College Hospital NHS Trust (Other); University Hospitals Sussex NHS Foundation (Unknown); Homerton University Hospital (Unknown); Barts & The London NHS Trust (Other); The Whittington Hospital NHS Trust (Other Government); Guy's and St Thomas' NHS Foundation Trust (Other); West Hertfordshire Hospitals NHS Trust (Other); Kingston Hospital NHS Trust (Other); Royal Free Hospital NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Epsom and St Helier University Hospitals NHS Trust (Other); Lewisham and Greenwich NHS Trust (Other Government); St George's University Hospital NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: EDGE 124858; IRAS 264198 (Other: Health Research Authority (HRA))
Record Dates: First submitted 2022-04-20; First posted 2022-05-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Pregnancy Related
Keywords: LGBTQIA+ Reproduction; Resilience; Vulnerability; Risk; Neonatal Health; Parent Health; Allostatic Load

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gestational parents: The study is composed of a sample of LGBTQIA+ and cisgender, heterosexual parents who are receiving antenatal care at the participating hospitals.

SUMMARY:
Pregnancy care typically assumes patients are heterosexual married women whose gender matches their assigned sex (i.e., cisgender), stigmatizing patients and creating limitations, blocking affirming care. Consequently, lesbian, gay, bisexual, queer, intersex, asexual, and/or transgender (LGBTQIA+) parents face minority stress as discrimination in antenatal care. This mixed-methods study assesses stressors and resilience factors on pregnancy and birth outcomes. LGBTQIA+ pregnant parents (n=200) are case-matched with cisheterosexual peers (n=600). Primary data comes from two panel surveys, one antenatally and one postpartum, combined with medical records. A sub-sample (n=30) will complete a journal between surveys. Findings will inform care guidelines and provider training.

DETAILED DESCRIPTION:
Patients using reproductive health services, like care during pregnancy (called antenatal care), are most often assumed to be heterosexual married women whose gender matched their sex assigned at birth (i.e., cisgender). Due to these assumptions, pregnancy care procedures are based on a sweeping assumption of who becomes pregnant and gives birth. This assumption is based on the pregnant person's gender and/or sexual orientation. As a result of this assumption, parents who are lesbian, gay, bisexual, queer, intersex, asexual, non-binary, and/or transgender (LGBTQIA+) can experience stress in the form of stigma, prejudice, and discrimination (i.e. "minority stress"). In the United Kingdom, there are 525,000 LGBTQIA+ potential gestational patients who may face this type of stress while receiving pregnancy care. That means that there is a preventable higher risk for pregnancy and birth complications caused by increased stress during pregnancy and daily life. These complications include macrosomia, pre-term birth, and low-birth weight. Preventable stress, also called minority stress, links to this increase in health problems outside of pregnancy as well. Since minority stress influences patient/parents' health, it is also called a risk or vulnerability. Resilience, or the ability to overcome stress and discrimination, can sometimes help improve health outcomes. However, little is known about which types of resilience can be helpful for LGBTQIA+ parents given their unique experiences of minority stress.

The planned observational study will investigate the ways in which experiences of minority stress and resilience in pregnancy care are associated with parent health and birth outcomes. A sample of pregnant patients (N=800) from maternity wards in and around London will take part through an online panel survey (completed twice) that will be linked to each patient/participant's electronic health records to create a quantitative dataset. Participant recruitment will focus on LGBTQIA+ pregnant patients (n=200). A matched comparison sample of cisgender, heterosexual pregnant patients (n=600) will also be recruited to take part from the same maternity. From the full sample, patient/parents from University College London Hospital will be invited to complete an at-home journal activity which will provide qualitative data on their experiences of minority stress and resilience. This smaller group (n=30). Results from this study can be used to inform LGBTQIA+ guidelines, training, and help make reproductive healthcare more inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Legal adult of reproductive age (18-49)
* Identifies as a lesbian, gay, bisexual, queer, nonbinary, intersex, and/or transgender (or cisgender and heterosexual for comparison sample)
* Currently pregnant and receiving antenatal care at one of the study sites

Exclusion Criteria:

* Any pregnant persons under the age of 18
* Pregnant individuals using sites locations for Urgent care, A&E, non-antenatal services only

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant people of all genders are welcome to participate within the study as long as they are receiving antenatal care at a participating Hospital Trust.
Study Population: Gestational parents receiving antenatal care in Greater London.
Sampling Method: Non-Probability Sample
Enrollment: 945 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Primary Scientific Aim - Parental Health | through study completion, up to 10 months
  The outcome measured for impact from resilience and vulnerability is parent health as allostatic load (as health data from routine antenatal check-ups). Scales will be composited into intrapersonal stressors (i.e., felt stigma, level of outness), interpersonal stressors (i.e., homelessness & child welfare, stressful life events/stress, everyday discrimination, chronic strains, police interactions), structural stressors (i.e., household social vulnerability index, deprivation score), intrapersonal resilience (i.e., coping, social support), interpersonal resilience (i.e., patient experience scale, shared decision-making, emotional reactivity), and structural resilience (i.e., community connectedness, civic engagement).
Primary Scientific Aim - Infant Health | through study completion, up to 10 months
  The composite for parent health (i.e. allostatic load from Outcome 1) will be assessed to see if there is an impact on infant health (a composite of head circumference, gestational length, birth weight, birth length, Apgar score).

SECONDARY OUTCOMES:
Secondary Scientific Aim - Understanding additional stressors and resilience | through study completion, up to 10 months
  Qualitative journals will be used to assess for additional stressors and resilience resources to ascertain if there are measures that have not been accounted for within the quantitative measures. These are presently unknown, as the point of the measure is to uncover these dimensions of the constructs of resilience and vulnerability.
Secondary Scientific Aim - Contextualising resilience and vulnerability | through study completion, up to 10 months
  The same qualitative journals in outcome 3 will also provided narratives about the experiences of parents with extreme resilience and vulnerability scores. The assessment of these narratives will be done to help contextualise the presence of extreme scores for parents receiving antenatal care at UCLH. The contents of these narratives collectively will be reported within the final findings alongside the quantitative data, as well as will be quoted specifically when relevant.

CONTACTS AND LOCATIONS:
Overall Officials: David M Frost, PhD, Study Chair — University College, London
Locations (14):
- United Kingdom (14):
  - King's College Hospital NHS Foundation Trust, Brixton
  - Kingston Hospital NHS Foundation Trust, Kingston upon Thames
  - Barts Health NHS Trust, London
  - Homerton University Hospital NHS Foundation Trust, London
  - Whittington Health NHS Trust, London
  - Royal Free London NHS Foundation Trust, London
  - Lewisham and Greenwich NHS Trust, London
  - St George's University Hospitals NHS foundation Trust, London
  - University College London Hospital NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Epsom and St Helier University Hospitals NHS Trust, Sutton
  - West Hertfordshire Teaching Hospitals NHS Trust, Watford
  - University Hospitals Sussex NHS Foundation, Worthing

IPD SHARING:
Plan to Share IPD: Undecided